CLINICAL TRIAL: NCT03791710
Title: Effect of Autologous Fat Grafting and Nanofat Usage on Burn Wound Healing and Early Scarring
Brief Title: Effect of Autologous Fat Grafting on Acute Burn Wound Healing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahmed Mohamed Abouzaid (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Abouzaid, specialist plastic, reconstructive surgery and burn therapy, Abouqir General Hospital
Organization: Abouqir General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbouqirBurn1
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Lipectomy; Floderm topical cream; Bandages; Skin Transplantation

STUDY DESIGN:
Intervention Model Description: two groups one will have the fat grafting and the other will be the control group treated with the conventional methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): this group of patients are treated with the regular conventional methods like application of topical agents e.g silver sulphadiazine
  Interventions: Drug: Topical Cream; Procedure: split thickness skin grafting
- fat grafting group (Active Comparator): this group of patients will have the autologous fat grafting for their burn wounds
  Interventions: Procedure: autologous fat grafting; Procedure: split thickness skin grafting

INTERVENTIONS:
Procedure: autologous fat grafting — regular liposuction procedure at which sufficient amount of fat is extracted from the patient and then the fat is processed then grafted underneath the burn wound
  Other Names: liposuction and lipofilling
  Arms: fat grafting group
Drug: Topical Cream — serial dressing with topical agents e.g Silver Sulphadiazine
  Other Names: dressing
  Arms: control group
Procedure: split thickness skin grafting — depridment and split thickness skin grafting
  Other Names: skin grafting

SUMMARY:
the study evaluates the role of autologous fat grafting and the usage of nanofat in the treatment of the acute burn injuries in different genders and its influences on the healing time and hospital stay, pain control, the need and take of a split thickness skin graft and its size, and the end resulting early scarring, in comparison with control group that were treated with traditional methods, so as to find out new method of treating burn injuries and decreasing its morbidity.

DETAILED DESCRIPTION:
as the patient is admitted, full evaluation locally ( as regard the wound itself and the areas of fat harvesting) and generally (assessment of the general condition) is done, fluid resuscitation is started as the unit protocol hand in hand with the analgesia and other medications prescribed according to the unit protocol.

the patient's general condition is optimized for surgery of the fat extraction and grafting which typically should be within the first 6 days of admission.

then under anesthesia (any possible type from local and regional up to general anesthesia) liposuction procedure is performed, then fat is processed then grafted at the wound site with other portion prepared as nanofat for topical use and wound coverage, then sterile dressing is applied.

typically follow up is held daily with the dressing change day after another with the use of the nanofat only and sterile dressing

ELIGIBILITY:
Inclusion Criteria:

* both males and females within the age frame are candidates.
* previously healthy individuals with no co-morbid conditions e.g cardiac, hepatic, diabetic, vascular or renal disease.
* with TBSA of 10 to 30% affected and of deep dermal to full thickness wound depth, at any part of the body except the genitalia, perineum or the perianal region or those with inhalational injury.

Exclusion Criteria:

* other patients aged younger or older than the specified age group.
* patients with co-morbid conditions.
* patients with smaller or larger BSA than the specified BSA.
* burns involving the genitalia, perineum or the perianal region and patients with inhalational injury.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
wound healing time | one to three weeks
  the effect of the fat grafting on the wound healing time

SECONDARY OUTCOMES:
effect on pain perception, subjective assessment scale | immediate post-operative and up to three weeks
  effect of the fat grafting on the pain sensation in the burn wound, assessment through a numerical scale starting at "0" indicating no pain at all to "10" the most intense severe pain. the range between "1" and "3" describes mild pain, between "4" and "6" describes moderate pain, and lastly from "7" to "10" severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abouzaid, MSc, Principal Investigator — Abouqir GH
Locations (1):
- Abouqir General Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abouzaid AM, El Mokadem ME, Aboubakr AK, Kassem MA, Al Shora AK, Solaiman A. Effect of autologous fat transfer in acute burn wound management: A randomized controlled study. Burns. 2022 Sep;48(6):1368-1385. doi: 10.1016/j.burns.2021.10.011. Epub 2021 Nov 1. PMID 34906386